CLINICAL TRIAL: NCT01750125
Title: Validation of Pulse Wave Doppler Demodulation Algorithm for the Continuous, Non-invasive Measurement of Blood Flow Velocity
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 16305
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Focus is on Healthy Subjects
Keywords: Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy subjects: In these health subjects we will measure ascending aortic blood flow with pulse wave Doppler and also record the raw audio of the Doppler signal
  Interventions: Device: measure ascending aortic blood flow with pulse wave Doppler

INTERVENTIONS:
Device: measure ascending aortic blood flow with pulse wave Doppler

SUMMARY:
The investigators hypothesize that performance of fast-Fourier transformation on the raw Doppler signals obtained from ascending aortic blood flow will recreate the pulse wave Doppler trace visualized on modern echocardiography machines, and that this will allow for the measurement and recording of vascular flow waveforms

DETAILED DESCRIPTION:
Currently there is no commercially available mechanism for the measurement of blood flow velocity waveforms non-invasively. Blood flow velocity waveforms require the use of invasive catheters, thus precluding clinical use. Such information would allow the researcher / practitioner the ability to continuously measure blood flow, pulse pressure, and the pulsatility index of any vascular structure accessible by ultrasound with minimal additional risk to the subject / patient. This data, when combined with arterial blood pressure data, could also be used to measure peripheral pressure volume loops as well as aortic vascular impedance, both of which cannot be currently measured in vivo.

The ability to measure blood flow velocity waveforms at high temporal resolution would provide clinicians with new tools for hemodynamic optimization (both a novel means of estimating myocardial oxygen consumption [pressure volume area] as well as afterload [aortic vascular impedance]) and researchers with the ability to conduct hemodynamic experiments that were not previously possible. This work will serve as the foundation for several other related projects which depend on the ability to continuously record blood flow velocity waveforms.

ELIGIBILITY:
Inclusion Criteria:

* 18-65
* Healthy

Exclusion Criteria:

* Cannot visualize ascending aorta with ultrasound

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects 18-65
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Comparison between estimated arterial flow waveform and pulse wave Doppler trace | day of procedure
  Estimated arterial flow waveform using fast Fourier transformation (FFT) will be compared to the pulse wave Doppler trace from the device

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States